CLINICAL TRIAL: NCT00953186
Title: Hyperbaric Oxygen Therapy as Adjunctive Treatment in Diabetics With Chronic Foot Ulcers
Brief Title: Hyperbaric Oxygen Therapy as Adjunctive Treatment of Chronic Diabetic Foot Ulcers
Acronym: HODFU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mrs. Thelma Zoegas Foundation (Other)
Collaborators: Lund University (Other); Region Skåne Sweden (Other Government); Gorthons Foundation Helsingborg Sweden (Unknown)
Responsible Party: Magnus Löndahl, MD, Senior consultant, Dept Endocrinology, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z012094
Record Dates: First submitted 2009-07-28; First posted 2009-08-06 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes; Foot Ulcer; Healing
Keywords: Diabetes; Foot ulcer; Neuropathy; Ischemia
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBOT (Active Comparator): 100 % oxygen at 2,5 atmospheres for 90 minutes/day, 5 days a week for 8 weeks
  Interventions: Device: HBOT
- Placebo (Placebo Comparator): air at 2,5 atmospheres for 90 minutes/day, 5 days a week for 8 weeks
  Interventions: Device: hyperbaric air

INTERVENTIONS:
Device: hyperbaric air — air at 2,5 atmospheres for 90 minutes/day, 5 days a week for 8 weeks treatment given in hyperbaric chamber
  Arms: Placebo
Device: HBOT — 100 % oxygen at 2,5 atmospheres for 90 minutes/day, 5 days a week for 8 weeks treatment given in hyperbaric chamber
  Arms: HBOT

SUMMARY:
The purpose of this study is to evaluate if hyperbaric oxygen therapy heels more foot ulcers as compared to placebo in patients with diabetes mellitus and chronic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus,
* foot ulcer with duration > 3 months,
* treatment at Diabetes foot clinic for > 2 months,
* vascular surgical intervention had not been recommended for the affected lower limb.

Exclusion Criteria:

* severe obstructive pulmonary disease,
* malignancy and untreated thyrotoxicosis),
* current drug or alcohol misuse,
* vascular surgery in the lower limbs within the last two months,
* participation in another study or suspected poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2002-06; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Ulcer healing | 3, 6, 9, 12, 18, 24 months

SECONDARY OUTCOMES:
Amputationrate | 6, 12, 24 months
time to ulcer healing | 24 months
QoL | 3, 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Löndahl, MD, Principal Investigator — Inst Clinical Sciences in Lund, Lund University, Sweden; Per L Katzman, ass prof, MD, Study Chair — Inst Clinical Sciences in Lund, Lund University, Sweden
Locations (1):
- Dept Anesthesiology, Helsingborg Hospital, Helsingborg, Sweden

REFERENCES:
- [Background] Londahl M, Katzman P, Nilsson A, Hammarlund C, Sellman A, Wykman A, Hugo-Persson M, Apelqvist J. A prospective study: hyperbaric oxygen therapy in diabetics with chronic foot ulcers. J Wound Care. 2006 Nov;15(10):457-9. doi: 10.12968/jowc.2006.15.10.26970. PMID 17124820
- [Derived] Londahl M, Katzman P, Hammarlund C, Nilsson A, Landin-Olsson M. Relationship between ulcer healing after hyperbaric oxygen therapy and transcutaneous oximetry, toe blood pressure and ankle-brachial index in patients with diabetes and chronic foot ulcers. Diabetologia. 2011 Jan;54(1):65-8. doi: 10.1007/s00125-010-1946-y. Epub 2010 Oct 19. PMID 20957342
- [Derived] Londahl M, Katzman P, Nilsson A, Hammarlund C. Hyperbaric oxygen therapy facilitates healing of chronic foot ulcers in patients with diabetes. Diabetes Care. 2010 May;33(5):998-1003. doi: 10.2337/dc09-1754. PMID 20427683